CLINICAL TRIAL: NCT00359385
Title: The Effects of Alendronate After Cure of Primary Hyperparathyroidism
Acronym: AlenPostPara
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: incomplete enrollment
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAB8202
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Hyperparathyroidism
Keywords: primary hyperparathyroidism; hyperparathyroidism; PHPT; PTH; hypercalcemia; bone density; osteoporosis; bone turnover; DXA; pQCT; cQCT; alendronate; Fosamax; parathyroid hormone; parathyroid surgery; parathyroidectomy; Silverberg; Rubin; Bilezikian; treatment
MeSH Terms: conditions — Hyperparathyroidism; Hyperparathyroidism, Primary; Hypercalcemia; Osteoporosis | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alendronate 70mg weekly (Active Comparator): Alendronate 70mg weekly
  Interventions: Drug: Alendronate 70mg weekly
- placebo of alendronate 70mg weekly (Placebo Comparator): placebo of Alendronate 70mg weekly
  Interventions: Drug: Alendronate 70mg weekly

INTERVENTIONS:
Drug: Alendronate 70mg weekly — 70mg weekly
  Other Names: Fosamax

SUMMARY:
We are investigating whether, after surgical cure of primary hyperparathyroidism, alendronate provides even greater beneficial skeletal effects than parathyroidectomy alone.

Primary Hyperparathyroidism (PHPT) is a disorder that can be associated with bone loss. After successful surgery for PHPT bone density improves without any treatment. However, it is possible that bone density might improve to an even greater extent if Fosamax is used after the surgical cure. Fosamax is approved by the FDA for the prevention and treatment of osteoporosis, and the goal of this project is to determine whether after successful surgical cure of PHPT, Fosamax is even better for the skeleton than just parathyroid surgery alone.

DETAILED DESCRIPTION:
Study Purpose:

Hypothesis: After successful surgical cure of primary hyperparathyroidism alendronate provides even greater beneficial skeletal effects than parathyroidectomy alone.

Primary hyperparathyroidism (PHPT) is typically a disorder of mild hypercalcemia. Skeletal involvement can be demonstrated when bone densitometry is performed. Effects of excess PTH on bone include preferential involvement of cortical bone (e.g. forearm) and relative sparing of cancellous bone (e.g. vertebral spine). Bone properties, such as bone turnover, size and geometry, are also altered in PHPT. The only cure for PHPT is removal of abnormal parathyroid tissue. In the absence of medical intervention, bone mass increases briskly after successful surgical treatment of PHPT. Parathyroid surgery also promptly reduces bone remodeling, typically increased in PHPT, to normal values. Bone resorption markers fall first, followed by bone formation markers. The difference in time course between the rapid fall in resorption markers and the more gradual fall in formation markers provides a window of time when bone mass increases rapidly. The post-surgical increase in BMD is attributed to a filling-in, or mineralization, of the enlarged, PTH-driven, remodeling space. Whether further gains in bone density could be achieved with more prompt and greater suppression of bone resorption in the postoperative period is unknown. The potent bisphosphonate, alendronate (Fosamax), reduces bone remodeling and enhances secondary mineralization. It has been shown to increase bone density in subjects with PHPT who do not undergo parathyroid surgery. The goal of this project is to test the hypothesis that after successful surgical cure of PHPT, alendronate provides even greater beneficial skeletal effects than parathyroidectomy alone.

Study Design and Statistical Analysis:

The clinical investigation will have as its primary outcome variable an increase in lumbar spine density (DXA) when alendronate is used during the first year after surgery. The patients will be stratified by BMD upon presentation, because we have shown a variable response to parathyroidectomy depending on initial spine BMD. The study design is a randomized, double-blind, placebo, 1-year, controlled clinical trial, in which patients will receive alendronate 70 mg weekly or a placebo tablet identical in appearance. As a secondary endpoint, we also plan to examine the effects of alendronate after parathyroidectomy on bone structure and skeletal dynamics using sensitive, state-of-the-art, non-invasive quantitative tools. With central and peripheral quantitative computed tomography, we will investigate changes in bone size, geometry and cortical porosity in cancellous and cortical bone. With serum and urinary markers of bone turnover, we will determine whether alendronate hastens control of bone resorption, thus enhancing the discordance between bone formation and resorption and leading to even greater improvements in bone mineral density.

There are 3 Specific Aims; all measurable after successful parathyroid surgery:

Specific Aim #1 to investigate the effects of alendronate on bone mineral density.

Specific Aim #2 to determine whether alendronate alters bone turnover to maximize the augmented window defined by a rapid fall in bone resorption and a slower fall in bone formation.

Specific Aim #3 to characterize the effects of alendronate on bone size and bone geometry in the cancellous and cortical skeletal compartments using QCT and pQCT

In Specific Aim #1 we will obtain the data for our primary outcome. This will include data regarding changes at the lumbar spine, as well as at the hip and distal 1/3 radius. The rate of change in BMD at these sites will also be determined by BMD measurements within the 1-year period of observation.

Specific Aim #2 will examine the potential mechanism for the greater improvements with bone density, namely a change in bone turnover dynamics that would favor greater accumulation of bone mineral with alendronate therapy.

With Specific Aim #3 we will obtain more detailed information about changes in bone structure that are likely to occur with more sophisticated tools than DXA. This will allow for specific assessment of changes in cancellous vs. cortical bone and in bone size, geometry and porosity.

Two groups of 20 patients each will self-administer a weekly oral pill, of alendronate or placebo, for 12 months. This number will give us the statistical power to make the observations that are planned. 18 subjects per group (n=36) allows detection of a between group difference of 0.059 gm/cm2 in lumbar spine BMD at one year, with a power of 80%, using a t-test and two-tailed alpha of 0.05. Calculation is based on our preliminary data in which bone density improves 0.053 ± 0.061 gm/cm2 (6.7% change) without intervention after surgery. We will be able to detect an overall change in treatment group of 0.053 + .059 = .112 gm/cm2, or 14% after surgery. We will recruit an additional 4 subjects (36+ 4 = 40) to account for drop-outs.

When the main publication has been published, or within two years from the completion of data collection, we will prepare a data sharing file that comprises the following components and accompanying annotation: the protocol, procedures manual, operations manual, blank copies of all report forms used in the study, the schedule of assessments, the data dictionary providing data storage specifications for each field, the study database tables representing the captured and audited data; the final data analytic data tables and the listing of the programming statements responsible for any data recoding or sub-setting, data summaries of each data table including descriptive statistics for validation of value integrity, and written description of the study conduct and noteworthy details anticipated to potentially affect data interpretation.

Study visits and Procedures:

Certain tests will be performed as part of accepted procedures in patients with PHPT, but most will be obtained specifically for research purposes.

There will be a total of 6 visits in the study: The pre-parathyroidectomy baseline/safety visit ("-1Month" visit) which will occur approximately one month prior to parathyroidectomy, and the post-parathyroidectomy baseline ("Zero visit") where they will begin study drug. There will also be a one-month ("M1"), three-month ("M3"), six-month ("M6"), and the twelve-month visit ("12M").

The "-1Month" visit:

At this visit, potential participants will be screened into the study. That is, consent will be obtained, inclusion and exclusion criteria will be satisfied, and baseline values will be obtained.

The testing that will be performed at this visit is divided into two categories: research and safety.

Research Testing includes DXA, QCT, and pQCT as well as serum and urinary indices of bone mineral metabolism (serum Calcium, PO4, Albumin, PTH, Vitamin D, P1NP, BSAP, and urinary NTX and DPD). This reflects the standard baseline information captured prior to parathyroidectomy in the clinical setting, which includes serum calcium, vitamin D, and PTH as well as bone mineral density by DXA.

Safety Testing includes the lab tests being performed to satisfy inclusion and exclusion criteria. From the participants pre-surgical testing for their parathyroidectomy (which will always include CBC, BMET, PT, PTT) we will be able to obtain baseline safety data. Other baseline safety tests we will obtain are serum BUN, Creatinine, AST and ALT.

The complete list of results being sought at the "-1Month" visit are:

Serum BUN, Creatinine, AST, ALT, Calcium, PTH, Vitamin D, PO4, Albumin, P1NP, BSAP and urinary NTX and DPD, as well as bone mineral density by DXA, QCT, and pQCT.

The "ZERO" visit:

In order to determine that parathyroidectomy is successful persons having this surgery routinely have a serum Calcium and PTH performed. The results of the serum Calcium in particular can immediately reflect the success of the surgery. Therefore, as a final screening criteria, participants will provide us with the results of their routine post-parathyroidectomy serum Calcium (and PTH, but that can be at a later time).

Study drug will be initiated no longer than one month after parathyroidectomy, since the changes in mineral metabolism will likely start immediately after surgery.

At this visit we will obtain serum Calcium and PTH for research purposes. We will also randomize participants at this visit to receive either alendronate or placebo of alendronate. We will provide participants with their study pills and they will take their first on the day following the ZERO visit.

The complete list of things being done at the "ZERO visit":

Serum Calcium and PTH

MONTH 1 visit:

Serum and urinary indices of bone mineral metabolism (serum Calcium, PO4, Albumin, PTH, Vitamin D, P1NP, BSAP, and urinary NTX and DPD) will be collected.

MONTH 3 visit:

Serum and urinary indices of bone mineral metabolism (serum Calcium, PO4, Albumin, PTH, Vitamin D, P1NP, BSAP, and urinary NTX and DPD) will be collected.

MONTH 6 visit:

Serum and urinary indices of bone mineral metabolism (serum Calcium, PO4, Albumin, PTH, Vitamin D, P1NP, BSAP, and urinary NTX and DPD) will be collected and DXA will be performed. Also, participants will be supplied with more study pills.

MONTH 12 visit:

Serum BUN, Creatinine, AST, ALT, Calcium, PTH, Vitamin D, PO4, Albumin, P1NP, BSAP and urinary NTX and DPD, as well as bone mineral density by DXA, QCT, and pQCT will be performed at this visit.

Study Drugs:

Alendronate, the study drug, has been shown to be very safe in many large, randomized, placebo-controlled trials in individuals with osteoporosis and is FDA- approved for prevention and treatment of osteoporosis. It has also been shown to be safe in individuals with PHPT. In clinical practice, the most common side effect with alendronate is gastrointestinal discomfort (for more information see RISKS). Study patients will be instructed about how to administer the alendronate (or placebo) so as to minimize the likelihood of this side effect.

Medical Devices:

Dual x-ray absorptometry (DXA), XtremeCT (pQCT), and QCT (cQCT)

ELIGIBILITY:
Inclusion Criteria:

* patients with PHPT who have a negative T-score by BMD at the lumbar spine before surgery;
* successful surgery for PHPT as documented by normalization of serum calcium and PTH levels within 1 week of study initiation.

Exclusion Criteria:

* vitamin D deficiency;
* any concomitant disease that might affect mineral metabolism such as hyperthyroidism, Paget's disease of bone, diabetes mellitus, chronic liver or renal disease, acromegaly, Cushing's syndrome, rheumatoid arthritis, myeloma;
* any woman who is within 5 years of the menopause;
* gastrointestinal disorders, surgery or drugs affecting absorption;
* treatment with a bisphosphonate within 2 years of parathyroidectomy;
* treatment with any of the following medications more recently than 6 months prior to enrollment: estrogens, progestins, raloxifene, calcitonin, systemic corticosteroids, fluoride, lithium, loop diuretics, methotrexate;
* abnormalities of the esophagus which delay esophageal emptying such as stricture or achalasia;
* inability to stand or sit upright for at least 30 minutes;
* increased risk of aspiration;
* hypersensitivity to alendronate;
* hypocalcemia;
* pregnancy or nursing; (women within childbearing years will be advised not to conceive during the study);
* age < 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To investigate the effects of alendronate on bone mineral density using data on changes at the lumbar spine, the hip and distal 1/3 radius. The rate of change in BMD at these sites will also be determined by BMD. | July 2009

SECONDARY OUTCOMES:
We also intend to determine whether alendronate alters bone turnover to maximize the augmented window defined by a rapid fall in bone resorption and a slower fall in bone formation. | July 2009

CONTACTS AND LOCATIONS:
Overall Officials: Shonni J. Silverberg, MD, Principal Investigator — Columbia University
Locations (1):
- CUMC, New York, New York, United States